CLINICAL TRIAL: NCT03335449
Title: Effects on Respiratory Mechanics of Two Different Ventilation Strategies During Robotic-Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPINAZZOLA GIORGIA (Other)
Responsible Party: Sponsor-Investigator, SPINAZZOLA GIORGIA, Physician, specialist in Anesthesia and Intensive Care Medicine, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 10398/14
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Mechanics; Mechanical Ventilation Complication

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protective ventilation group (Experimental): Protective ventilation (PV group) (Vt 6 ml/Kg of ideal body weight, PEEP 8-10 cmH 2 O and repeated recruitment maneuvers.
  Interventions: Other: Protective ventilation group
- Standard ventilation group (No Intervention): Standard ventilation (SV group) (Tidal Volume, Vt 10 ml/Kg of ideal body weight, Positive End Expiratory Pressure, PEEP 5 cmH 2 O, no recruitment maneuvers)

INTERVENTIONS:
Other: Protective ventilation group — Application of a protective ventilation strategy in order to improve gas exchange and respiratory mechanics during Robotic surgery in deep Trendelenburg position.
  Other Names: Low tidal volume, high PEEP and recruitment maneuvers
  Arms: Protective ventilation group

SUMMARY:
This Randomized controlled clinical study, entitled "Effects on Respiratory mechanics of two different ventilation strategies during Robotic- Gynecological surgery", is an original paper. The study was performed in Rome, Italy, from September 2014 to September 2015.

Nowadays several studies evaluated the effects of "open lung strategy" and the positive effect of Recruitment Maneuvers and Positive End Expiratory Pressure (PEEP) application during general anesthesia, especially during open abdominal surgery and in elderly patients.

This is the first study aimed at evaluating two different ventilation strategies in healthy respiratory women undergoing Robotic surgery. In particular, the investigators evaluated the effects of protective ventilation strategy on respiratory mechanics, gas exchange and post-operative respiratory complications compared to standard ventilation.

DETAILED DESCRIPTION:
The ventilation protocol consisted in volume-controlled mechanical ventilation through Ventilator, inspiratory to expiratory ratio of 1:2, and a respiratory rate adjusted to normocapnia (end-tidal carbon dioxide partial pressure between 30 and 40 mmHg). The were randomly assigned to Standard (SV) or Protective (PV) group.

participants in the SV group received a Tidal Volume (Vt) of 10 ml/kg of Ideal Body Weight (IBW) and a PEEP of 5 cmH2O, the participants in the PV group a Vt of 6 ml/kg of IBW and a PEEP of 8-10 cmH2O, associated to recruitment maneuvers (RMs).

RMs were performed only in hemodynamic stable conditions and at pre-set moments: after the induction of anesthesia, after any disconnection from the mechanical ventilator, each hour during the surgical procedures and immediately before extubation. RMs were performed in Pressure Control mode as follows: the limit of peak inspiratory pressure was set at 45 cmH2O and the pressure control was set at 30 cmH2O, therefore three consecutive thirty seconds lasting inspiratory pauses were performed. At the end of RMs, respiratory rate, inspiratory to expiratory ratio, inspiratory pause, and Vt were set back at values preceding the RMs.

Air Flow (V') was measured with a heated pneumotachograph, inserted between the Y-piece of the ventilator circuit and the endotracheal tube. The pneumotachograph was linear over the experimental range of flow. Volume was obtained by numerical integration of the flow signal. Airway pressure (Paw) was measured proximal to the endotracheal tube with a pressure transducer with a differential pressure of ± 100 cm H2O. The end-inspiratory and end-expiratory occlusions were performed through specific maneuver of ventilator.

Following end-inspiratory occlusion there is an immediate drop of the airway pressure from a maximal value (Pmax) to airway pressure at zero flow (P1), followed by a further decrease to plateau pressure (P2). The plateau pressure usually arrived within 3 seconds. Therefore, airway pressure 3 seconds after occlusion was taken as the static end-inspiratory elastic recoil pressure (P2) of the respiratory system. The use of the interrupter method for the measurement of respiratory mechanics allows possible quantification of the airway and viscoelastic properties of the respiratory system. The difference between Pmax and P1 divided by flow provides major information about minimal airway resistance (Rmin), while the difference between P1 and P2 (ΔP) divided by flow stands for viscoelastic resistance or Pendelluft effect of the respiratory system (ΔR). Maximal respiratory resistance (Rmax) is the sum of Rmin and ΔR. The inspiratory volume divided by P2- Total PEEP yields respiratory system compliance. Mechanical respiratory measurements and arterial blood gases were performed immediately after intubation, after pneumoperitoneum (AP), every hour during the procedure and before extubation (Ext). A further arterial blood gas sample was analyzed 1 hour after extubation.

The day after the surgical procedure, clinical patient examination and chest x ray were performed, in order to detect eventual pulmonary adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Gynecological cancer elegible for laparoscopic surgery

Exclusion Criteria:

* Respiratory disease
* Obesity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Compliance | One year
  inspiratory Volume/Plateau Pressure-PEEP (ml/cmH2O)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Valenza F, Chevallard G, Fossali T, Salice V, Pizzocri M, Gattinoni L. Management of mechanical ventilation during laparoscopic surgery. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):227-41. doi: 10.1016/j.bpa.2010.02.002. PMID 20608559
- [Background] Fahy BG, Barnas GM, Flowers JL, Nagle SE, Njoku MJ. The effects of increased abdominal pressure on lung and chest wall mechanics during laparoscopic surgery. Anesth Analg. 1995 Oct;81(4):744-50. doi: 10.1097/00000539-199510000-00015. PMID 7574004
- [Background] Perilli V, Sollazzi L, Bozza P, Modesti C, Chierichini A, Tacchino RM, Ranieri R. The effects of the reverse trendelenburg position on respiratory mechanics and blood gases in morbidly obese patients during bariatric surgery. Anesth Analg. 2000 Dec;91(6):1520-5. doi: 10.1097/00000539-200012000-00041. PMID 11094011
- [Background] Maracaja-Neto LF, Vercosa N, Roncally AC, Giannella A, Bozza FA, Lessa MA. Beneficial effects of high positive end-expiratory pressure in lung respiratory mechanics during laparoscopic surgery. Acta Anaesthesiol Scand. 2009 Feb;53(2):210-7. doi: 10.1111/j.1399-6576.2008.01826.x. PMID 19175578
- [Background] Talab HF, Zabani IA, Abdelrahman HS, Bukhari WL, Mamoun I, Ashour MA, Sadeq BB, El Sayed SI. Intraoperative ventilatory strategies for prevention of pulmonary atelectasis in obese patients undergoing laparoscopic bariatric surgery. Anesth Analg. 2009 Nov;109(5):1511-6. doi: 10.1213/ANE.0b013e3181ba7945. PMID 19843790

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03335449/Prot_SAP_000.pdf